CLINICAL TRIAL: NCT06252662
Title: Liposomal Bupivacaine Vs Bupivacaine with Dexmedetomidine in an Erector Spinae Plane Block for Mastectomies in Cancer Patients: a Randomized Control Trial
Brief Title: Liposomal Bupivacaine Vs Bupivacaine with Dexmedetomidine in Erector Spinae Plane Blocks for Mastectomies
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Principal Investigator, Grant Miller, Chair Acute Pain Service Anesthesia Department, Principal Investigator, Clinical Professor, United States Naval Medical Center, Portsmouth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-18229
Record Dates: First submitted 2024-01-31; First posted 2024-02-12 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: erector spinae plane block; bupivacaine; morphine equivalents; pain score; post-operative pain; post-surgical pain; liposomal bupivacaine; Exparel
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: single blinded randomized control trial.
Who Masked: Participant
Masking Description: Patients will not be able to see overhear from the block team the type of drugs used in the block.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal bupivacaine and bupivacaine plain erector spinae plane block (Active Comparator): Erector spinae plane block performed on the surgical side (left, right or bilateral) as appropriate based on planned surgical consent. Utilizing ultrasound to see the fascial layers and guide the needle placement under direct visualization. Block will include 1.33% liposomal bupivacaine 10ml plus 0.25% bupivacaine plain 20 ml per side of the block.
  Interventions: Drug: Liposomal bupivacaine
- Bupivacaine plain with dexmedetomidine (Experimental): Erector spinae plane block performed on the surgical side (left, right or bilateral) as appropriate based on planned surgical consent. Utilizing ultrasound to see the fascial layers and guide the needle placement under direct visualization. Block will include 0.25% bupivacaine plain 30 ml plus dexmedetomidine 0.5 mcg/kg per side of the block.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — block duration extension additive
  Other Names: Precedex
  Arms: Bupivacaine plain with dexmedetomidine
Drug: Liposomal bupivacaine — Control arm, comparison for block duration with dexmedetomidine
  Other Names: Exparel
  Arms: Liposomal bupivacaine and bupivacaine plain erector spinae plane block

SUMMARY:
Perform a comparison of effective pain relief duration between liposomal bupivacaine and dexmedetomidine when added to bupivacaine in a block for mastectomy for cancer surgery. The erector spinae plane block is a well-established block that is utilized for post operative pain control for procedures performed on the soft tissue of the chest and chest wall as well as intrathoracic procedures. The goal is comparison of the effective duration of both study groups to determine if there is a significant difference in time and amount of post operative opioids required which admitted to hospital.

DETAILED DESCRIPTION:
Performance of a single-blinded randomized control trial to evaluate effectiveness of postoperative pain control in erector spinae plane blocks with bupivacaine with liposomal bupivacaine as the control versus bupivacaine with dexmedetomidine. Plan to randomize patients by alternating months, so that odd months' patients will receive bupivacaine 0.25% with liposomal bupivacaine in the erector spinae plane block. Even months patients will receive bupivacaine 0.25% with dexmedetomidine in the erector spinae plane block.

Block will be performed with ultrasound by the Acute Pain Service team. A time out confirming location of surgery, allergies, consents completed prior to start of the block. Patients will be monitored with 5 lead electrocardiography, non-invasive blood pressure, and pulse oximetry. After skin wheal with 1% lidocaine via 25-27 g needle and echogenic 20 g needle will be utilized to perform the block. The needle will be placed under direct ultrasound visualization into the erector spinae plane. The plane will be hydro dissected with normal saline to confirm needle tip has accessed the erector spinae plane. The local anesthetic will be given in a total of 0.2 ml/kg up to 20 mls (selected based on the study group placement) and aspiration will occur every 5 mls during the block. This will be repeated on the second side if a bilateral block is indicated in based on the surgical consent. All patients will receive 10 mg IV dexamethasone post-induction of anesthesia.

While the patient is in patient pain scores and milligrams of morphine equivalence (MMEs) will be collected every 6 hours based on charting by the nurses providing care starting from time "0" in the PACU after surgery, up until discharge. Then to obtain pain scores up to 72 hours after surgery, patients will be called at home after 72 hours and asked what their pain scores had been daily since discharge and a total of tabs taken daily.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring any variation of mastectomy with or without axillary lymph node dissection.
* Patient agrees to a peripheral nerve block.
* Patient agrees to be a study participant.
* APS team believes a peripheral nerve block would be appropriate for the patient after reviewing medical/surgical history.
* Surgeon agrees with the block plan by APS.

Exclusion Criteria:

* Patient declines a peripheral nerve block.
* Patient declines to be a study participant.
* APS team believes a peripheral nerve block is not clinically indicated.
* Surgeon does not want a peripheral nerve block.
* Patient has allergy to local anesthestic.
* Patient has an active infection at the site of the peripheral nerve block.
* Patient with pre-existing neural deficits along the distribution of the block.
* Patient with coagulopathy.
* Patient taking antithrombotic drugs outside the ASRA guidelines.
* Patients weight is less that 50 kg due to concerns for local anesthetic toxicity syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Is bupivacaine with dexmedetomidine superior to liposomal bupivacaine in both density and duration? | 96 hours
  Control group erector spinae plane block with liposomal bupivacaine is less dense and not as long lasting as bupivacaine with dexmedetomidine experimental group. Will investigate initial visual analog scale (VAS) pain scores to determine how effective the block is after surgery and every 6 hours while in patient. Additionally, calling the patient discharging after 96 hours from the time of the block and collect daily pain scores from the patient. This is to establish which group had best pain scores throughout and longest duration of lowest pain scores.

SECONDARY OUTCOMES:
Evaluate oral milligram of morphine equivalent (MME). | 96 hours
  Same control and experimental group assessing for morphine milligram equivalents reduction between groups. Will investigate milligram of morphine equivalent every 6 hours to see how much each group requires. In particular looking for increasing trend in morphine equivalence over time. Additionally, calling the patient discharging after 96 hours from the time of the block and collect daily opioid medications taken by the patient and converting to milligram morphine equivalents. This is to establish which group has taken the least amount of morphine equivalents throughout the duration of the block, as an indication to the duration of optimum benefit of the block.

OTHER OUTCOMES:
Time to first opioid administration | 24 hours
  Determine if there is a difference in time to first opioid dose after surgery when block is provided before surgery. To determine if there is a difference in the quality of the block after the surgery requiring earlier administration of opioids, as is expected with less dense block having more increased pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Haddock NT, Garza R, Boyle CE, Liu Y, Teotia SS. Defining Enhanced Recovery Pathway with or without Liposomal Bupivacaine in DIEP Flap Breast Reconstruction. Plast Reconstr Surg. 2021 Nov 1;148(5):948-957. doi: 10.1097/PRS.0000000000008409. PMID 34705768
- [Background] Schnabel A, Reichl SU, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of paravertebral blocks in breast surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2010 Dec;105(6):842-52. doi: 10.1093/bja/aeq265. Epub 2010 Oct 14. PMID 20947592
- [Background] Leong RW, Tan ESJ, Wong SN, Tan KH, Liu CW. Efficacy of erector spinae plane block for analgesia in breast surgery: a systematic review and meta-analysis. Anaesthesia. 2021 Mar;76(3):404-413. doi: 10.1111/anae.15164. Epub 2020 Jul 1. PMID 32609389
- [Background] Brown CA, Ghanouni A, Williams R, Payne SH, Ghareeb PA. Safety and Efficacy of Liposomal Bupivacaine Supraclavicular Nerve Blocks in Open Treatment of Distal Radius Fractures: A Perioperative Pain Management Protocol. Ann Plast Surg. 2023 Jun 1;90(6S Suppl 4):S332-S336. doi: 10.1097/SAP.0000000000003464. Epub 2023 Jan 31. PMID 36752544
- [Background] Malan SH, Jaroszewski DE, Craner RC, Weis RA, Murray AW, Meinhardt JR, Girardo ME, Abdelrazek AS, Borah BJ, Dholakia R, Smith BB. Erector Spinae Plane Block With Liposomal Bupivacaine: Analgesic Adjunct in Adult Pectus Surgery. J Surg Res. 2023 Sep;289:171-181. doi: 10.1016/j.jss.2023.03.016. Epub 2023 Apr 28. PMID 37121043
- [Background] Fidkowski CW, Choksi N, Alsaden MR. A randomized-controlled trial comparing liposomal bupivacaine, plain bupivacaine, and the mixture of liposomal bupivacaine and plain bupivacaine in transversus abdominus plane block for postoperative analgesia for open abdominal hysterectomies. Can J Anaesth. 2021 Jun;68(6):773-781. doi: 10.1007/s12630-020-01911-1. Epub 2021 Jan 11. PMID 33432496
- [Background] Nguyen A, Grape S, Gobbetti M, Albrecht E. The postoperative analgesic efficacy of liposomal bupivacaine versus long-acting local anaesthetics for peripheral nerve and field blocks: A systematic review and meta-analysis, with trial sequential analysis. Eur J Anaesthesiol. 2023 Sep 1;40(9):624-635. doi: 10.1097/EJA.0000000000001833. Epub 2023 Apr 10. PMID 37038770
- [Background] Kim DH, Liu J, Beathe JC, Lin Y, Wetmore DS, Kim SJ, Haskins SC, Garvin S, Oxendine JA, Ho MC, Allen AA, Popovic M, Gbaje E, Wu CL, Memtsoudis SG. Interscalene Brachial Plexus Block with Liposomal Bupivacaine versus Standard Bupivacaine with Perineural Dexamethasone: A Noninferiority Trial. Anesthesiology. 2022 Mar 1;136(3):434-447. doi: 10.1097/ALN.0000000000004111. PMID 35041742
- [Background] Albrecht E, Vorobeichik L, Jacot-Guillarmod A, Fournier N, Abdallah FW. Dexamethasone Is Superior to Dexmedetomidine as a Perineural Adjunct for Supraclavicular Brachial Plexus Block: Systematic Review and Indirect Meta-analysis. Anesth Analg. 2019 Mar;128(3):543-554. doi: 10.1213/ANE.0000000000003860. PMID 30303864
- [Background] Abdallah FW, Brull R. Facilitatory effects of perineural dexmedetomidine on neuraxial and peripheral nerve block: a systematic review and meta-analysis. Br J Anaesth. 2013 Jun;110(6):915-25. doi: 10.1093/bja/aet066. Epub 2013 Apr 15. PMID 23587874
- [Background] Pehora C, Pearson AM, Kaushal A, Crawford MW, Johnston B. Dexamethasone as an adjuvant to peripheral nerve block. Cochrane Database Syst Rev. 2017 Nov 9;11(11):CD011770. doi: 10.1002/14651858.CD011770.pub2. PMID 29121400